CLINICAL TRIAL: NCT04732533
Title: Feasibility of Home-based tES for Older Adults at Risk of Falling
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-16; Pro00044339 (Other: Advarra IRB)
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Aging; Accidental Falls
Keywords: Mobility; Dual Task
MeSH Terms: interventions — TES; Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Single group, open-label intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tES (transcranial electrical stimulation) (Experimental): All participants in phase 1 received the tDCS (transcranial direct current stimulation) intervention. For each new potential participant recruited into Phase 2, 3 or 4, the type of tES intervention, either tDCS or a combination of tDCS and tACS (transcranial alternating current stimulation) will be determined at the discretion of the study PI in consultation with the participant.
  The tDCS intervention will be administered with the goal of facilitating the excitability of the left dlPFC (dorsolateral prefrontal cortex).
  The combination of tDCS and tACS intervention will be administered with the goals of 1) using tDCS to facilitate the excitability of the left dlPFC using the parameters outlined in the preceding paragraph, and at the same time, 2) using tACS targeting the left angular gyrus at gamma frequency 40 Hz.
  Interventions: Other: tES (transcranial electrical stimulation)

INTERVENTIONS:
Other: tES (transcranial electrical stimulation) — Phase 1: The participant will receive 10, 20-minute sessions of tDCS on Monday-Friday, at approximately the same time of day, over two consecutive weeks.
  Phase 2: The participant will receive 22, 20-minute sessions of tES. 10 sessions will take place over the first two weeks on Monday-Friday, at approximately the same time of day. This will be followed by 3 tES sessions per week over four weeks.
  Phase 3: The participant will receive up to 260, 20-minute sessions of tES. The participant can complete up to 5 tDCS sessions per week over 52 weeks.
  Phase 4: The participant will receive up to 780, 20-minute sessions of tES. The participant can complete up to 5 tDCS sessions per week over 156 weeks.

SUMMARY:
In this project, the investigators propose to demonstrate the feasibility of remotely-monitored, caregiver (or spouse)-administered, home-based tES (transcranial electrical stimulation) intervention to improve mobility in ambulatory older adults with recent falls. This is a four-phase feasibility study in older, ambulatory adult participants at risk of falling due to a loss of balance (participant faller, PF) together with a willing and able participant administrator (PA) that is available during weekdays to administer tES to the PF.

Phase 1 is focused on the development and refinement of our training materials for home-based tDCS (transcranial direct current stimulation) for PF/PA pairs. The objectives of this phase:

1. Identify areas of confusion and challenges for older adults.
2. Refine our training materials to accompany the home-based tDCS system.

In Phase 2, the investigators will complete a pilot trial in 12 PF/PA pairs to assess the feasibility of deploying home-based tES in larger clinical trials, and to prepare for the development and implementation of such trials. The objectives of this phase:

1. Determine the mean/range number of visits needed for in-person training.
2. Compliance and retention with the study protocol.
3. Safety/side effects of home-based tES, as compared to previously established laboratory-based tES data.

The investigators hypothesize that adult PAs are able to successfully administer home-based tES to PFs. The investigators also expect that PF/PA pairs will exhibit excellent adherence to the intervention and that the prevalence and severity of reported tDCS side-effects will be similar to that observed in previous laboratory-based studies.

In Phase 3, the investigators will complete a pilot trial in up to 18 PF/PA pairs; i.e., those who have previously successfully completed either Phase 1 or Phase 2. The study objectives/aims for Phase 3 are:

1. Further explore compliance and retention with the study protocol over a longer time period
2. Identify safety/side effects of home-based tES over a longer time-period as compared to previously established laboratory-based tDCS interventions.

In Phase 3, the investigators hypothesize that adult PA's who have previously demonstrated the ability to successfully administer tES at home, will retain competence and compliance with administration over a longer period, up to 1 year.

In Phase 4, we will complete a pilot trial in up to 18 PF/PA teams; those who have previously successfully completed Phase 3. The study objective/aims for Phase 4 will be to:

1. Identify Safety, effectiveness and adherence to home-based tES over longer period of time as compared to previously established laboratory-based tES interventions.
2. Further explore the proof of Concept for the home-based tES interventions

In Phase 4 we hypothesize that adult PA's who have previously demonstrated the ability to successfully administer tES at home, will adhere with the study protocol over a longer period of time, up to 3 years.

DETAILED DESCRIPTION:
In older adults, falls are costly, consequential and correlated with both physical and cognitive decline. Most falls occur when standing or walking, especially when completing these tasks in complex environments or while simultaneously performing additional cognitive tasks. To this end, older adults with worse cognitive "executive" function have worse mobility and are more likely to fall.

Transcranial Electrical Stimulation (tES), which includes both transcranial Direct Current Stimulation (tDCS) and transcranial Alternating Current Stimulation (tACS), holds promise as a therapy to improve dual task standing and walking and other "high-level" aspects of mobility in older adults. tES is a low cost technique, is very safe with only minimal side effects, is portable and is very easy to administer. However, tES must be administered numerous times per week for several consecutive weeks in order to induce lasting therapeutic benefit. As each tES session must currently be administered in clinical or laboratory settings, such interventions are not currently available to many older adults--especially those who 1) live far away from the clinical/laboratory, and/or 2) have physical and/or cognitive limitations that make it difficult to organize and utilize transportation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will be the same for PF/PA pairs in both Phase 1 and Phase 2 of the study. All participant pairs who complete either Phase 1 or 2 will be eligible to complete Phase 3. All participant teams who complete Phase 3 in its entirety will be eligible to complete Phase 4

PF group:

* Aged 60+
* Self-report of one or more falls within the past year, and/or concern of falling in the future, and/or self-report of Parkinson's disease.
* Able to read, write, and communicate in English
* Able to identify an eligible PA to participate with them in the study

PA group:

* At least 21 years of age
* Able to read, write, and communicate in English
* Self-reported computer proficiency and willingness to learn how to use tDCS
* Stated availability during weekdays throughout the study period to administer tDCS to the PF

Exclusion Criteria:

* Exclusion criteria will be the same for PF/PA pairs in both Phase 1 and Phase 2 of the study.

PF group:

* Evidence of cognitive impairment that would likely interfere with one's ability to understand the study protocol, risks/benefits, and testing procedures. This will be defined as self-reported diagnosis of Alzheimer's disease or dementia, a score of ≤19 on the Telephone Interview for Cognitive Status (TICS) at the time of telephone screening, a score of 18 or less on the Montreal Cognitive Assessment (MoCA) during the in-person screen, or an inability to understand study procedures following review of the Informed Consent form.
* Inability to stand or ambulate unassisted for at least 25 feet.
* Contraindications to tDCS, including a reported seizure within the past two years, use of neuro-active drugs, the risk of metal objects in the brain, skull, or head, self-reported presence of specific implanted medical devices (e.g., deep brain stimulator, medication infusion pump, cochlear implant), or the presence of any active, uncontrolled dermatological condition, such as eczema, on the scalp.

PA group:

* Mild cognitive impairment defined by a TICS score ≤34 during the phone screen, a MoCA score ≤24 during the in-person screen, or insufficient understanding of study procedures following review of the Informed Consent form.
* Poor eyesight, severe arthritis in the hands, pain, deformity or other condition that interferes with successful administration of tDCS.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Screening to enrollment ratio ("percent", 0-100, higher ratio means a better outcome) | The whole data collection period of phase 2 (~ 6 weeks for the whole study)
  The number of screenings needed to enroll one participant
Intervention adherence rate ("percent", 0-100, higher ratio means a better outcome) | The whole data collection period (~ 6 weeks for phase 2; ~ 52 weeks for phase 3; ~156 weeks for phase 4)
  Number of tDCS sessions completed
Side effects | The whole data collection period (~ 6 weeks for phase 2; ~ 52 weeks for phase 3; ~156 weeks for phase 4)
  The number, type, severity and duration of reported side effects
Training sessions | The whole data collection period (~ 6 weeks for phase 2; ~ 52 weeks for phase 3; ~156 weeks for phase 4)
  The number of training sessions needed for PAs to successfully and comfortably administer home-based tDCS

SECONDARY OUTCOMES:
Change from baseline in the dual task cost to gait speed (reduced dual task cost after intervention means a better outcome) | The whole data collection period (~ 6 weeks for phase 2; ~ 52 weeks for phase 3; ~156 weeks for phase 4)
  The change from baseline in the degree to which performing a secondary cognitive task diminishes gait speed
Change from baseline in the dual task cost to standing postural sway speed (reduced dual task cost after intervention means a better outcome) | Before and after the intervention (~ 6 weeks for phase 2; ~ 52 weeks for phase 3; ~156 weeks for phase 4)
  The change from baseline in the degree to which performing a secondary cognitive task diminishes the control of standing posture.
Change from baseline in Trail Making Test B - A (reduced time after intervention means a better outcome) | Before and after the intervention (~ 6 weeks for phase 2; ~ 52 weeks for phase 3; ~156 weeks for phase 4)
  The change from baseline in cognitive executive function
Change from baseline in gait speed (increased value after intervention means a better outcome) | Before and after the intervention (~ 6 weeks for phase 2; ~ 52 weeks for phase 3; ~156 weeks for phase 4)
  The change from baseline in gait speed
Change from baseline in Timed Up-and-Go (TUG) (reduced time after intervention means a better outcome) | Before and after the intervention (~ 6 weeks for phase 2; ~ 52 weeks for phase 3; ~156 weeks for phase 4)
  The change from baseline in overall mobility function
Change from baseline in Montreal Cognitive Assessment (MoCA) total score (increased score after intervention means a better outcome) | Before and after the intervention (~ 6 weeks for phase 2; ~ 52 weeks for phase 3; ~156 weeks for phase 4)
  The change from baseline in global cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Brad Manor, PhD, Principal Investigator — Hebrew SeniorLife
Locations (1):
- Hebrew Rehabilitation Center, Roslindale, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The HSL Institute for Aging Research will promote the development of new research and new investigators by making the data available to outside investigators. The database will include longitudinal demographic, clinical, functional, and physiologic from all participants.
  All data will be stripped of primary identifiers and entered into a master database. All data collection procedures, variable definitions and codes, field locations, and frequencies will be documented in a separate file.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The investigators will make the data and associated documentation available once summary data are published or otherwise made available, starting six months after publication.
Access Criteria: The investigators will make the data and associated documentation available to users only under a data-sharing agreement that provides for: 1) a commitment to using data only for research purposes and not to identify any particular participant; 2) a commitment to securing the data using appropriate computer technology; and 3) a commitment to destroying or returning the data after analyses are completed. The availability of data will be advertised over the Internet through websites maintained by Hebrew SeniorLife and Harvard Medical School.
  All investigators wishing to access the data will submit a brief proposal describing their research project, data needs, regulatory approvals, and mechanisms to assure patient confidentiality. Upon affirmative review by the Principal Investigator and co-investigators of this study, a data-sharing agreement will be signed and the requesting investigators will be given a working data file and appropriate documentation.